CLINICAL TRIAL: NCT01331512
Title: The InChianti Follow-Up Study
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903320; 03-AG-N320
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-02

CONDITIONS: Aging; Decrease in Ambulation
Keywords: Clinical Geriatrics; Biomechanics; Epidemiology; Decline in Ambulation

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Older persons are often referred to physicians because of mobility difficulties that grow worse as they age. To better understand the reasons for mobility difficulties in older persons, researchers conducted a population-based study of individuals living in the Chianti geographic area of Tuscany, Italy. Researchers are now interested in conducting a follow-up study on the original participants to assess the effects of aging on their mobility.

Objectives:

- To conduct a follow-up study on the participants in the mobility study of older persons in the Greve in Chianti and Bagno a Ripoli areas near Florence, Italy.

Eligibility:

- Original participants in the InChianti Mobility Study.

Design:

* The InChianti Follow-up Study will repeat most elements of the baseline evaluation from the original study. Participants will be seen on the 3-year anniversary of their baseline study assessment.
* Participants will have a home interview with questions about their physical and mental health, family history, daily activities, and living conditions related to their continued mobility.
* Participants will provide blood and urine samples, and will have tests of heart and motor nerve function and imaging studies of bones and the circulatory system.
* Participants will also have a functional evaluation of their motor skills, including walking tests, range of motion tests, and grip strength.

DETAILED DESCRIPTION:
In the past decade epidemiologic and clinical studies have described the prevalence and incidence of disability and have elucidated demographic characteristics, health behaviors, diseases, and physiologic impairments that are associated with increased risk of developing disability in old age. Mobility disability has emerged as a critical aspect of functioning. Mobility, defined as the ability to move independently from one point to another, is a critical part of maintaining independence and an essential attribute of quality of life. In those age 85 years and older, nearly 60 percent of women and 40 percent of men have difficulty walking two to three blocks. Older people who are mobile are more likely to remain in the community, have lower rates of subsequent morbidity and mortality, and have higher quality of life. Recent work in biomechanics, clinical geriatrics, epidemiology, and clinical trials has helped to improve our understanding of the decline in walking ability in old age and the influence of multiple intrinsic and extrinsic factors. However, a great deal is still not understood about how older persons progressively lose the ability to ambulate. The InChianti Study has the potential to make major new advances in our knowledge of progressive decline in ambulation in older persons.

A great deal of information is available from the baseline evaluation in this study and the crosssectional analyses that can be done with these data will be very valuable. There are, however, limitations in what we can learn from cross-sectional data. The baseline data revealed many relationships between factors that were studied and disability, but there may be circularity in these relationships that cannot be sorted out if we only have cross-sectional data available. For example, abnormalities in certain biomarkers may be a cause of disability or may be caused by disability. Only by doing longitudinal analyses that begin with non-disabled persons can the temporal sequence be determined. Cross-sectional analyses only permit the study of factors that are currently related to disability while longitudinal analyses allow for the identification of subclinical markers of risk that predict future disability onset. There is therefore much to be gained by performing a follow-up evaluation of the cohort to obtain longitudinal data.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 65 years and older

Must reside in Greve in Chianti or Bagno A Ripoli, Italy

Subjects with modertative cognitive problems will be included as long as the consent can be read and signed by by a first-degree relative of the participant or, in absence of first-degree relative, another relative living with or close to the participant

EXCLUSION CRITERIA:

Children

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1167 (Actual)
Dates: Start 2003-01-31; Study Completion 2015-01-02

CONTACTS AND LOCATIONS:
Overall Officials: Tamara B Harris, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Research and Care on Aging, Florence, Italy

REFERENCES:
- [Derived] Pellegrino R, Paganelli R, Di Iorio A, Bandinelli S, Mussi C, Sparvieri E, Volpato S, Tanaka T, Ferrucci L. Lack of Immune Resilience Negatively Affects Physical Resilience: Results From the InCHIANTI Follow-Up Study. J Gerontol A Biol Sci Med Sci. 2024 May 1;79(5):glae076. doi: 10.1093/gerona/glae076. PMID 38457361
- [Derived] Hidalgo-Liberona N, Merono T, Zamora-Ros R, Rabassa M, Semba R, Tanaka T, Bandinelli S, Ferrucci L, Andres-Lacueva C, Cherubini A. Adherence to the Mediterranean diet assessed by a novel dietary biomarker score and mortality in older adults: the InCHIANTI cohort study. BMC Med. 2021 Nov 24;19(1):280. doi: 10.1186/s12916-021-02154-7. PMID 34814922
- [Derived] Cattelani L, Palumbo P, Palmerini L, Bandinelli S, Becker C, Chesani F, Chiari L. FRAT-up, a Web-based fall-risk assessment tool for elderly people living in the community. J Med Internet Res. 2015 Feb 18;17(2):e41. doi: 10.2196/jmir.4064. PMID 25693419
- [Derived] Dashti HS, Follis JL, Smith CE, Tanaka T, Cade BE, Gottlieb DJ, Hruby A, Jacques PF, Lamon-Fava S, Richardson K, Saxena R, Scheer FA, Kovanen L, Bartz TM, Perala MM, Jonsson A, Frazier-Wood AC, Kalafati IP, Mikkila V, Partonen T, Lemaitre RN, Lahti J, Hernandez DG, Toft U, Johnson WC, Kanoni S, Raitakari OT, Perola M, Psaty BM, Ferrucci L, Grarup N, Highland HM, Rallidis L, Kahonen M, Havulinna AS, Siscovick DS, Raikkonen K, Jorgensen T, Rotter JI, Deloukas P, Viikari JS, Mozaffarian D, Linneberg A, Seppala I, Hansen T, Salomaa V, Gharib SA, Eriksson JG, Bandinelli S, Pedersen O, Rich SS, Dedoussis G, Lehtimaki T, Ordovas JM. Habitual sleep duration is associated with BMI and macronutrient intake and may be modified by CLOCK genetic variants. Am J Clin Nutr. 2015 Jan;101(1):135-43. doi: 10.3945/ajcn.114.095026. Epub 2014 Nov 26. PMID 25527757
- [Derived] Tanaka T, Ngwa JS, van Rooij FJ, Zillikens MC, Wojczynski MK, Frazier-Wood AC, Houston DK, Kanoni S, Lemaitre RN, Luan J, Mikkila V, Renstrom F, Sonestedt E, Zhao JH, Chu AY, Qi L, Chasman DI, de Oliveira Otto MC, Dhurandhar EJ, Feitosa MF, Johansson I, Khaw KT, Lohman KK, Manichaikul A, McKeown NM, Mozaffarian D, Singleton A, Stirrups K, Viikari J, Ye Z, Bandinelli S, Barroso I, Deloukas P, Forouhi NG, Hofman A, Liu Y, Lyytikainen LP, North KE, Dimitriou M, Hallmans G, Kahonen M, Langenberg C, Ordovas JM, Uitterlinden AG, Hu FB, Kalafati IP, Raitakari O, Franco OH, Johnson A, Emilsson V, Schrack JA, Semba RD, Siscovick DS, Arnett DK, Borecki IB, Franks PW, Kritchevsky SB, Lehtimaki T, Loos RJ, Orho-Melander M, Rotter JI, Wareham NJ, Witteman JC, Ferrucci L, Dedoussis G, Cupples LA, Nettleton JA. Genome-wide meta-analysis of observational studies shows common genetic variants associated with macronutrient intake. Am J Clin Nutr. 2013 Jun;97(6):1395-402. doi: 10.3945/ajcn.112.052183. Epub 2013 May 1. PMID 23636237